CLINICAL TRIAL: NCT02327416
Title: A Prospective Randomized Clinical Trial of Combination Sequential Treatment With Y Peginterferon Alfa-2b and ETV (Entecavir) in CHB (Chronic Hepatitis B) Patients NAs (Nucleotides or Nucleosides) Experienced (Anchor Study)
Brief Title: A Prospective Clinical Trial in Chronic Hepatitis B Patients NAs (Nucleotides or Nucleosides) Experienced (Anchor Study)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Qin Ning, Director and Chair of Department of Infectious Diseases, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Anchor study
Record Dates: First submitted 2014-11-23; First posted 2014-12-30 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2b; Colony-Stimulating Factors; entecavir; adefovir dipivoxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1,conventional control group (Active Comparator): Drug: Entecavir and or adefovir dipivoxil are used for 96 weeks and the follow up 24 weeks. Entecavir 0.5mg po daily or plus ADV （adefovir dipivoxil）10mg po daily.
  Interventions: Drug: Entecavir and or adefovir dipivoxil
- 2，combination and sequential group (Experimental): Drug: Y peginterferon Alfa-2b 180 micrograms sc/week for 96 weeks; Drug: Entecavir and or adefovir dipivoxil are used for 48 weeks. Entecavir 0.5mg po daily for 48 weeks or plus ADV 10mg po daily.
  Interventions: Drug: Y peginterferon alfa-2b; Drug: Entecavir and or adefovir dipivoxil
- 3, multitarget group (Experimental): Drug: Y peginterferon Alfa-2b 180 micrograms sc/week for 96 weeks; Drug: Granulocyte-macrophage colony stimulating factor is used for 48 weeks; Drug: Entecavir and or adefovir dipivoxil are used for 48 weeks. Entecavir 0.5mg po daily for 48 weeks or plus ADV 10mg po daily.
  Interventions: Drug: Y peginterferon alfa-2b; Drug: Granulocyte-macrophage colony stimulating factor; Drug: Entecavir and or adefovir dipivoxil

INTERVENTIONS:
Drug: Y peginterferon alfa-2b — In arm 2 and 3, Y peginterferon alfa-2b is used for 96 weeks
  Other Names: peginterferon alfa-2b
  Arms: 2，combination and sequential group; 3, multitarget group
Drug: Granulocyte-macrophage colony stimulating factor — In arm 3, Granulocyte-macrophage colony stimulating factor is used for 48 weeks intermittently
  Other Names: GMCSF
  Arms: 3, multitarget group
Drug: Entecavir and or adefovir dipivoxil — In arm 1, Entecavir and or adefovir dipivoxil are used for 96 weeks and the follow up 24 weeks as conventional control, In arm 2 and 3, Entecavir and or adefovir dipivoxil are used for 48 weeks.
  Other Names: ETV and or ADV

SUMMARY:
This study is a multi-center, randomized, prospective, open-label Phase III Clinical trial to assess the efficacy and safety of combination and sequential treatment with Y peginterferon Alfa-2b,entecavir and GMCSF in chronic hepatitis B patients nucleotides or nucleosides experienced. Patients were randomized to one of 3 groups to receive different antiviral treatment.

DETAILED DESCRIPTION:
Patients who have been pretreated with and responded to one or two nucleotides or nucleosides for at least one year, with HBV (Hepatitis B Virus) DNA less than 1000 copies/ml and HBsAg less 3000 IU/ml were randomized to one of 3 groups, to receive Y peginterferon Alfa-2b 180mcg/week for 96 weeks, entecavir 0.5 mg po daily for 48 weeks plus GMCSF (Granulocyte-macrophage colony stimulating factor) for 48 weeks, or Y peginterferon Alfa-2b 180mcg/week for 96 weeks and entecavir 0.5 mg po daily for 48 weeks, or only ETV for 96 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients from 18 to 65 years of age;
2. HBsAg positive, entecavir and or adefovir dipivoxil are used at least 1 year including patients with nucleotides or nucleoside resistance history if their HBV DNA obtained control;
3. Before nucleotides or nucleosides treatment, ALT > 2 ULN, HBV DNA >10000 copies/ml,HBsAg positive;
4. Serum HBV DNA < 1000 copies/ml;
5. Serum HBsAg < 3000 IU/ml;
6. HBsAg positive;
7. Negative urine or serum pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of test drug;
8. Absence of cirrhosis confirmed by ultrasonic test;
9. Agree to participate in the study and sign the patient informed consent.

Exclusion Criteria:

1. Patients who had NAs resistance and HBV DNA > 1000 copies/ml, or treatment of drugs with IFN longer than 6 months;
2. Other antiviral, anti-neoplastic or immunomodulatory treatment (including supra physiologic doses of steroids and radiation) 6 months prior to the first dose of randomized treatment (except for 7 days of acyclovir for herpetic lesions more than 1 month prior to first administration of randomized treatment). Patients who are expected to need systemic antiviral therapy other than that provided by the study at any time during their participation are also excluded;
3. Women with ongoing pregnancy or breast-feeding;
4. Co-infection with active hepatitis A, hepatitis C, hepatitis D(Those hospitals which have the ability to do the test will do) and/or human immunodeficiency virus (HIV);
5. ALT >10 ULN;
6. Evidence of decompensated liver disease (Child-Pugh score > 5 ). Child-Pugh > 5 means, if one of the following 5 conditions are met, the patient has to be excluded:

   one of the following 5 conditions are met, the patient has to be excluded:
   1. Serum albumin < 3.5 g/L;
   2. Prothrombin time > 3 seconds prolonged;
   3. Serum bilirubin > 34 µ mol/L;
   4. History of encephalopathy;
   5. History of variceal bleeding;
   6. Ascites;
7. History or other evidence of a medical condition associated with chronic liver disease other than viral hepatitis (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures, thalassemia);
8. Signs or symptoms of hepatocellular carcinoma, patients with a value of alpha-fetoprotein > 100 ng/mL are excluded, unless stability (less than 10% increase) has been documented over at least the previous 3 months. Patients with values < 20 ng/mL but > 100 ng/mL may be enrolled, if hepatic neoplasia has been excluded by liver imaging;
9. Neutrophil count < 1500 cells/mm3 or platelet count <90,000 cells/mm3 at screening;
10. Hemoglobin < 11.5 g/dL for females and <12.5 g/dL for men;
11. Serum creatinine level > 1.5 ULN in screening period.
12. Phosphorus < 0.65 mmol/L;
13. ANA > 1:100;
14. History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquilizer at therapeutic doses for major depression or psychosis, respectively, for at least 3 months at any previous time or any history of the following: a suicidal attempt hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease;
15. History of a severe seizure disorder or current anticonvulsant use;
16. History of immunologically mediated disease, (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, rheumatoid arthritis etc.);
17. History of chronic pulmonary disease associated with functional limitation;
18. Diseases that IFN and Nucleotides or nucleosides are not suitable.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-10; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of HBsAg loss at week 96 | week 96
  Change from baseline in Percentage of HBsAg loss at week 96

SECONDARY OUTCOMES:
Change from baseline in HBsAg quantification and HBsAg decline at week 96 | week 96
  HBsAg quantification and HBsAg decline from baseline are measured.
Change from baseline in HBsAg seroconversion at week 96 | week 96
  HBsAg seroconversion from baseline is measured.

OTHER OUTCOMES:
Percentage of HBeAg loss or HBeAg seroconversion at week 96 for HBeAg positive patients | week 96
  Percentage of HBeAg loss or HBeAg seroconversion are measured at week 96 for patients with HBeAg positive at baseline
Percentage of HBV DNA normalization and ALT normalization at week 96 | week 96
  Percentage of HBV DNA normalization and ALT normalization at week 96 are measured.
Percentage of sustained virology response at week 120 | week 120
  Sustained virology response is measure at follow up week 24

CONTACTS AND LOCATIONS:
Overall Officials: Qin Ning, Doctor, Principal Investigator — Department of Infectious Diseases, Tongji Hospital
Locations (4):
- China (4):
  - Beijing Youan Hospital, Beijing, Beijing Municipality
  - Tongji Hospital, Wuhan, Hubei
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

REFERENCES:
- [Derived] Wu D, Huang D, Peng S, Chen Y, Yang F, Zhang X, Fu L, Xu L, Jiang J, Zheng Q, Chen X, Liu Y, Dou X, Ma K, Xi D, Wang P, Sun L, He R, Tian Y, Yin P, Yan W, Han M, Ning Q. Efficacy and safety of entecavir, peginterferon alfa-2b and GM-CSF combination therapy: the anchor randomized controlled trial. Hepatol Int. 2025 Dec 9. doi: 10.1007/s12072-025-10977-2. Online ahead of print. PMID 41366186
- [Derived] Gu M, Wu W, You J, Wu Q, Huang F, Zhang Y, Wang P, Xi D, Yan W, Wang X, Chen T, Wu D, Ning Q, Han M. High-Throughput Viral Integration Detection Reveals Baseline Breakpoints Burden Associated With HBsAg Seroclearance. Aliment Pharmacol Ther. 2025 Nov;62(9):887-900. doi: 10.1111/apt.70270. Epub 2025 Jul 16. PMID 40665748
- [Derived] Huang D, Wu D, Wang P, Wang Y, Yuan W, Hu D, Hu J, Wang Y, Tao R, Xiao F, Zhang X, Wang X, Han M, Luo X, Yan W, Ning Q. End-of-treatment HBcrAg and HBsAb levels identify durable functional cure after Peg-IFN-based therapy in patients with CHB. J Hepatol. 2022 Jul;77(1):42-54. doi: 10.1016/j.jhep.2022.01.021. Epub 2022 Feb 8. PMID 35149125